CLINICAL TRIAL: NCT06313697
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose Administration of GR2102 Injection in Healthy Adult Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Pharmacologic of GR2102
Brief Title: A Study to Evaluate the Safety, Immunogenicity, and Pharmacokinetics of GR2102 in Healthy Adult
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR2102-001
Record Dates: First submitted 2024-03-05; First posted 2024-03-15 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-03

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: respiratory syncytial virus; RSV; respiratory infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment group 1 (Experimental): single dose
  Interventions: Biological: GR2102 injection; Biological: placebo
- Treatment group 2 (Experimental): single dose
  Interventions: Biological: GR2102 injection; Biological: placebo
- Treatment group 3 (Experimental): single dose
  Interventions: Biological: GR2102 injection; Biological: placebo
- Treatment group 4 (Experimental): single dose
  Interventions: Biological: GR2102 injection; Biological: placebo
- Treatment group 5 (Experimental): single dose
  Interventions: Biological: GR2102 injection; Biological: placebo
- Treatment group 6 (Experimental): single dose
  Interventions: Biological: GR2102 injection; Biological: placebo

INTERVENTIONS:
Biological: GR2102 injection — single dose
Biological: placebo — single dose

SUMMARY:
the goal this clinical trail is to evaluate the safety、Pharmacokinetic and immunogenicity of GR2102 injection。 Subjects will be enrolled in different groups in sequential order, and within each group will be randomly assigned to receive either GR2102 injection or placebo administration, with each Subjects will be enrolled in only one of these groups。

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single-dose administration study to evaluate the safety, tolerability, pharmacokinetics, and preliminary pharmacodynamic profile of GR2102 Injection in healthy adult Chinese subjects.

After signing the informed consent form, subjects who meet the criteria for enrollment will be entered into different groups according to the randomization number.Subjects will be enrolled in only one of these groups.

Only after the 8 subjects in the current group have completed at least 7 days of safety and tolerability observations and have been determined to be safe and tolerable, will another group of subjects be allowed to proceed to the next group .

After completion of dosing, follow-up will be at least 150 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subjects
2. Signed informed consent

Exclusion Criteria:

1. Signs and symptoms of upper respiratory tract infection prior to randomization
2. Prior use of RSV vaccine or RSV antibody-based medications
3. history of malignant tumor

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-03-23 (Actual); Primary Completion 2025-01-06 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 150 days post dose
  to characterise the safety and tolerability of GR2102,including abnormal vital signs,laboratory tests,electrocardiogram and physical examination

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration | 150 days post dose
  Pharmacokinetic indices
Terminal Elimination Half Life | 150 days post dose
  Pharmacokinetic indices
anti-respiratory syncytial virus neutralizing antibodies titer levels | 150 days post dose
  indicator of immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: wei zhao, PHD, Principal Investigator — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No